CLINICAL TRIAL: NCT07207265
Title: Comic Relief: Graphic Medicine as Care for Caregivers
Status: Completed | Type: Observational
Sponsor: University of California, Riverside (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jennifer Syvertsen, Associate Professor Anthropology Department, University of California, Riverside
Other Study IDs: Comic Relief: Graphic Medicine; U54MD013368-05 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mental Wellbeing
Keywords: comics; art workshops; trauma; compassion fatigue; burnout
MeSH Terms: conditions — Wounds and Injuries; Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group intervention: weekly group sessions: Outcome measures:
  Skovholt Practitioner Professional Resiliency and Self-Care Inventory (Skovholt, 2010) ProQOL: Professional Quality of Life Screening (Stamm, 1997-2008)

SUMMARY:
Community care workers have been stretched to their capacity and exposed to ongoing trauma through their work addressing persistent health disparities in Inland Empire communities. The coronavirus pandemic and gap in Covid-19 mortality for minorities have highlighted the chronic stressors of racial injustice and dispossession that predate the pandemic and explain why these populations have higher comorbidities. While the pandemic has exacerbated ongoing stressors, the map of this crisis of care may show the way to deeper solutions. The premise of this project is that care occurs in a continuum of caretakers who also require care. The proposal seeks to address and complicate the question: who cares for the caregivers? This study will interrogate the benefits of providing a comics-making workshop, combined with trauma education and somatic experiencing, as a set of resiliency tools for care providers working with traumatized populations.

DETAILED DESCRIPTION:
The investigators will recruit up to 20 care workers from community-based organizations to participate in a series of comics workshops, who may also exhibit their work locally. The team will rigorously assess participants' experiences and changes in their wellbeing over time. This project provides preliminary data and a groundwork for larger investigations of how creating a space where caretakers can come together, learn about trauma healing and resiliency building, and share their post-traumatic growth and struggles with one another, increases both the resiliency of caretakers and the larger community.

ELIGIBILITY:
Inclusion Criteria:

18 years of age or more, Any care workers in the Inland Empire (Riverside or San Bernardino Counties) will be eligible to participate.

Exclusion Criteria:

There are no other specific exclusion criteria in terms of age, race, or gender, though we will aim to recruit a diverse sample that reflects the diversity in our community.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community care workers have been stretched to their capacity and exposed to ongoing trauma through their work addressing persistent health disparities in Inland Empire communities. The study is open to anyone living in the Riverside area who works a caregiver, broadly construed. This may include people working in education, healthcare, and non-profits.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Skovholt Practitioner Professional Resiliency and Self-Care Inventory | 1 art workshop per week for 7 weeks
  Skovholt Practitioner Professional Resiliency and Self-Care Inventory (Skovholt, 2010).
  * sub-scale professional vitality (range - 8-40)
  * sub-scale personal vitality (range - 11-55)
  * sub-scale professional stress (range - 9-45)
  * sub-scale personal stress. (range - 10-50) While there is no "optimal" score, higher scores on these scales indicate better outcomes or better ability to navigate stress.
ProQOL: Professional Quality of Life | 1 workshop per week for 7 weeks
  ProQOL: Professional Quality of Life Screening (Stamm, 1997-2008)
  * Compassion satisfaction is about the pleasure you derive from being able to do your work well. (avg score = 37)
  * Burnout is associated with feelings of hopelessness and difficulties in dealing with work or in doing your job effectively. (avg score = 22)
  * Compassion fatigue, also called secondary trauma and related to Vicarious Trauma, is about your work-related, secondary exposure to extremely stressful events.(avg score = 13) Higher scores on the compassion scale are better; lower scores on burnout and compassion indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Syvertsen, Principal Investigator — University of California, Riverside
Locations (1):
- University of Riverside, California, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: No
Because only 13 participants were enrolled in this pilot study, there is a heightened risk of identification even if direct identifiers are removed. Small sample sizes make it much easier for someone to infer or link data back to an individual based on combinations of demographics or clinical features. For these reasons, the Principal Investigator will not share the full individual-level dataset.

REFERENCES:
- See also: Graphic Medicine as Care for the Caregivers — https://www.carecooperativeie.com/blank